CLINICAL TRIAL: NCT01526915
Title: Contribution of Platelet Rich Fibrin (PRF) After Tooth Avulsion in the Prevention of Healing Delay and of Jawbone Osteochemonecrosis Induced by Bisphosphonates
Brief Title: Assessment of Platelet Rich Fibrin Efficiency on Healing Delay and on Jawbone Osteochemonecrosis Provoked by Bisphosphonates
Acronym: OCN/PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBM 2009-01; 2009-A01003-54 (Other: ID RCB - AFSSAPS)
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Jawbone Osteochemonecrosis Induced by Bisphosphonates
Keywords: PRF; PLATELET RICH FIBRIN; BISPHOSPHONATES
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone curettage + PRF (Experimental): Bone curettage and PRF insertion
  Interventions: Procedure: Bone curettage + PRF
- Bone curettage alone (Other): Bone curettage without PRF insertion
  Interventions: Procedure: Bone curettage alone

INTERVENTIONS:
Procedure: Bone curettage + PRF — Bone curettage and PRF insertion
  Arms: Bone curettage + PRF
Procedure: Bone curettage alone — Bone curettage without PRF insertion
  Arms: Bone curettage alone

SUMMARY:
The main objective of our study is to assess, after tooth extraction, the efficacity of PRF in the prevention of healing delay and of jawbone osteochemonecrosis induced by bisphosphonates

DETAILED DESCRIPTION:
Scientific Context Bisphosphonates (BP) work by slowing down bone remodelling. They are used in the management of different types of cancers and for the treatment of osteoporosis. Recent studies warned that this drug could produce adverse effects on jawbones .In December 2007, the AFSSAPS (French agency for the Sanitary Security of Health Products) alerted the health professionals about the risks of spontaneous or induced osteonecrosis following invasive odontological procedures on patients receiving BP. Prevalence of these osteonecrosis varies from 6% to 10% after surgical intervention. A healing delay estimated between 20 to 25% of cases frequently precedes the occurrence of osteochemonecrosis.

On the whole , the total rate of all complications amounts to 30%. We are extremely limited in terms of prevention or treatment of an OCN patient. We intend to study a biological autologous sediment obtained from a blood sample for its capacity to avoid these complications supervening. The collection of a coagulum called Platelet Rich Fibrin or PRF susceptible to provide the essential ingredients for the mucous membrane and the bone healing is obtained by centrifugation. This biomaterial rich in autologous fibrin is a concentrate of leukocytes, platelets and a number of factors favouring cicatrisation and immune response. Clinical applications are already well documented in orthopaedic, thoracic and cardiac surgeries and, also in dermatology. The use of PRF in dental surgery is more recent. Literature on this topic is very limited but these new techniques give rise to high hopes. Since February 2007,thanks to the classification as a medical treatment by the AFSSAPS, the PRF technique has been authorized.

Objectives To appraise after dental avulsion the PRF efficiency in preventing delay of cicatrisation and jawbone osteochemonecrosis induced by BP.

This efficiency will be assessed by a retroalveolar X-ray performed at each visit. The main criteria for evaluation is the discovery of cicatrisation delay at week 8 and/or osteochemonecrosis during the follow up.

Material and methods

Studied population: current or previous patients treated with BP and referred for a dental avulsion.

General experimental procedure: A prospective, longitudinal, multicentric, randomized open study. Patients will be randomized into two groups: dental avulsion only or dental avulsion and PRF. For both groups the initial management is surgical (bone curettage + PRF for the PRF group).The follow up is spread over one year with 10 visits. Each patient will undergo a clinical and photographic examination with a complete radiological check up(OPT),a standard biological blood test (blood count with haemogram (NFS) and a thorough calculation of the quantity of BP administered. The appearance of OCN or of any delay in cicatrisation will be documented by a histological biopsy, a bacteriological swab test and X-ray.

The requisite number of patients:

270 patients are required to validate the expected objectives in this study. Their recruitment will take place in 4 establishments: Metz-Thionville CHR (Regional Central Hospital) and three university teaching hospitals (CHU) Dijon, Nancy and Reims.

Total Duration of the study :

The estimated total duration will be 3 years: a 2 year recruitment with a 1 year follow-up.

Expected results and prospects To prove the interest of using PRF as a therapy able to prevent a delay in cicatrization or an OCN induced by BP.

ELIGIBILITY:
Inclusion Criteria:

* Patient major(male or female)
* Documented indication at the initial visit at day 0 (JO) for a maximum extraction of 3 teeth.
* Treatment with nitrogenous or non-nitrogenous BP by intravenous injection or oral administration whichever the reason for this drug prescription:

  * on going BP treatment
  * patient having received a previous treatment with bisphosphonates (irrespective of the duration and withdrawal date of this treatment)
* Patient having received the specific information letter regarding the study and having signed the clarified consent form.

Exclusion Criteria:

* Patient having a maxillary or mandibulary OCN at Day 0(JO)
* Positive HIV serology at Day 0(for patients belonging to the PRF group)
* Previous history of maxillo-cervico-facial radiotherapy
* Patients with estimated survival expectancy shorter than one year
* Lack of social security cover
* Inability of the patient to respect the study follow-up
* Patient having reached his/her majority and under tutelage,trusteeship or protection of the court
* Patient whose diagnosis could not be revealed to him/her (especially when the patient or their family expressed this wish).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Delay in cicatrisation at week 8 | 8 weeks
The appearance of osteochemonecrosis during the follow-up period | 1 year

SECONDARY OUTCOMES:
The characteristics of the received BP treatment: starting date of ongoing treatment, accumulated dose, type of BP, administration route | 1 year
The precise location of the extraction site according to the tooth classification number | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric GERARD, Dr, Principal Investigator — CHR Metz Thionville
Locations (5):
- France (5):
  - Chu de Dijon, Dijon
  - Scm Bally Curien, Maxéville
  - Chr Metz Thionville, Metz
  - Chu de Nancy, Nancy
  - Chu de Reims, Reims

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376